CLINICAL TRIAL: NCT05857306
Title: Effect of Olvanil Supplementation on Clinical, Biochemical and Anthropometric Parameters in Obese Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, ERIKA MARTINEZ-LOPEZ, Principal Investigator, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CI-01123
Record Dates: First submitted 2023-02-20; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Obesity
Keywords: Capsaicin analogs; Olvanil; Anthropometry
MeSH Terms: conditions — Obesity | interventions — olvanil

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Double-blind randomized parallel clinical trial
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator) Both types of capsules were made and packed in blisters and identical boxes. Every box was identified and tagged with a specific number by an associate researcher who is not involved in the recruitment, attention, or follow-up of the enrolled subjects.
  Finally, block randomization was the selected technique for this purpose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olvanil (Active Comparator)
  Interventions: Dietary Supplement: Olvanil
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Olvanil — Nutritional recommendation along with 4 mg Olvanil (1 capsule daily)
  Subects within the Intervention group will be provided with a nutritional recommendation along with Olvanil capsules. Subjects will be asked to consume one capsule per day. Every capsule contains: 4 mg Olvanil and 255 mg soy lecithin as excipient
  Arms: Olvanil
Dietary Supplement: Placebo — Nutritional recommendation along with 255 mg soy lecithin (1 capsule daily)
  Subects within the placebo group will be provided with a nutritional recommendation along with placebo capsules. Subjects will be asked to consume one capsule per day. Every capsule contains: 255 mg soy lecithin
  Arms: Placebo

SUMMARY:
Capsaicinoids are defined as alkaloid compounds of the Capsicum genus, they are characterised by the pungent flavor of chili. About the Capsicum genus, there are more than 20 known compounds, including dihydrocapsaicin, nordihydrocapsaicin, homodihydrocapsaicin and homocapsaicin. Capsaicin is the most popular compound in the biotechnological food industries. Recent studies has demonstrated the benefits of capsaicin in weight loss, however, the use of this molecule is limited given its high pungent capacity. Pungency develops due to the high affinity of capsaicin for the transient vanilloid potential receptor type 1 (TRPV1), which is primarily responsible for the transmission of pain. In order to eliminate pungency, capsaicin analogs have been developed, such as olvanil, this can become an alternative for its biotechnological and pharmaceutical purposes as an antiobesogenic treatment.

DETAILED DESCRIPTION:
A total of 56 subjects will be invited to be enrolled in a study approaching the properties of a capsaicin analog: olvanil, along with nutritional guidance.

This double blind, randomized, parallel clinical trial will consist in a 8-week intervention with recurrent visits every 4 weeks. In every visit, all subjects will undergo a body composition analysis as well as blood tests.

This study proposes three objectives for reaching a further understanding of the effects of olvanil:

1. Compare the anthropometric parameters at baseline versus final time between the groups.
2. Compare the clinical parameters at baseline versus final time between groups.
3. Compare the concentrations of the biochemical parameters at baseline versus final time between the groups.

Once the project is finished, the research strategies for new studies will be improved. In the same way, the application of the knowledge generated in it will be encouraged towards the health care of patients with obesity who could attend our service on future occasions. Finally, we would disseminate the knowledge generated in our institutional community, which would increase the impact of the project.

ELIGIBILITY:
Inclusion Criteria:

* 25-59 years of age
* Both sexes
* Subjects who agree to participate in the study and all signed informed consent
* BMI 30 kg/m2 - 39.9 kg/m2

Exclusion Criteria:

* Currently consuming any of the following drugs: NSAIDs, anticoagulants, hypoglycemic, oR hypolipemic drugs
* Diagnosed autoimmune diseases
* Diagnosed cancer
* Pregnancy and breastfeeding
* Suffering from gastritis and hemorrhoids
* Subjects who wish to abandon the study

Ages: 25 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Analysis of anthropometric variable (Height) | 8 weeks
  The measure will be performe without shoes, and an Height measurement will be determine by a stadiometer and represented in meters.
Analysis of anthropometric variable (Waist circumference) | 8 weeks
  The measure will be performe with light clothes. Waist circumference (WC) represented in centimeters was measured using a Lufkin Executive® Thinline 2-mm measuring tape.
Analysis of anthropometric variable (Body fat percentage) | 8 weeks
  The measure will be performe without shoes, with light clothes. Tetrapolar body electrical bioimpedance will be use to assess body fat percentage using InBody 370 and RJL Quantum V.
Analysis of anthropometric variable (Weight) | 8 weeks
  The measure will be performe without shoes, with light clothes and represented in kilograms Tetrapolar body electrical bioimpedance will be use to assess weight using InBody 370.
Analysis of anthropometric variable (BMI) | 8 weeks
  BMI will be calculate as weight in kilograms divided by height in square meters (kg/m2).
Analysis of clinic variables (Systolic and diastolic blood pressure) | 8 weeks
  The measurement of systolic and diastolic blood pressure will be carry out with a OMRON wireless upper arm blood pressure monitor, and represented millimeters of mercury (mmHg)
Analysis of biochemicals variables (Glucose) | 8 weeks
  Biochemical measurements at baseline and after 8 weeks supplementation Blood samples will be taken after 8 to 10 h of fasting and then centrifuged to obtain the serum, which will be frozen at -80 °C.
  - Glucose (Glu) mg/dL
  Will be carry out by dry chemistry using a Vitros 350 Analyzer.
Analysis of biochemicals variables (Triglycerides) | 8 weeks
  Biochemical measurements at baseline and after 8 weeks supplementation Blood samples will be taken after 8 to 10 h of fasting and then centrifuged to obtain the serum, which will be frozen at -80 °C.
  Determinations of:
  - Triglycerides (TG) mg/dL,
  Will be carry out by dry chemistry using a Vitros 350 Analyzer.
Analysis of biochemicals variables (Total cholesterol) | 8 weeks
  Biochemical measurements at baseline and after 8 weeks supplementation Blood samples will be taken after 8 to 10 h of fasting and then centrifuged to obtain the serum, which will be frozen at -80 °C.
  Determinations of:
  - Total cholesterol (TC) mg/dL,
  Will be carry out by dry chemistry using a Vitros 350 Analyzer.
Analysis of biochemicals variables (High-density lipoprotein) | 8 weeks
  Biochemical measurements at baseline and after 8 weeks supplementation Blood samples will be taken after 8 to 10 h of fasting and then centrifuged to obtain the serum, which will be frozen at -80 °C.
  Determinations of:
  - High-density lipoprotein (HDL) mg/dL,
  Will be carry out by dry chemistry using a Vitros 350 Analyzer.
Analysis of biochemicals variables (Low-density lipoprotein) | 8 weeks
  Biochemical measurements at baseline and after 8 weeks supplementation Blood samples will be taken after 8 to 10 h of fasting and then centrifuged to obtain the serum, which will be frozen at -80 °C.
  Determinations of:
  - Low-density lipoprotein (LDL) mg/dL,
  Will be carry out by dry chemistry using a Vitros 350 Analyzer.
Analysis of biochemicals variables (Very low-density lipoprotein) | 8 weeks
  Biochemical measurements at baseline and after 8 weeks supplementation Blood samples will be taken after 8 to 10 h of fasting and then centrifuged to obtain the serum, which will be frozen at -80 °C.
  Determinations of:
  - Very low-density lipoprotein (VLDL) mg/dL,
  will be carry out by dry chemistry using a Vitros 350 Analyzer.
Analysis of biochemicals variables (Creatinine) | 8 weeks
  Biochemical measurements at baseline and after 8 weeks supplementation Blood samples will be taken after 8 to 10 h of fasting and then centrifuged to obtain the serum, which will be frozen at -80 °C.
  Determinations of:
  - Creatinine (mg/dL),
  will be carry out by dry chemistry using a Vitros 350 Analyzer.
Analysis of biochemicals variables (Serum bilirubin) | 8 weeks
  Biochemical measurements at baseline and after 8 weeks supplementation Blood samples will be taken after 8 to 10 h of fasting and then centrifuged to obtain the serum, which will be frozen at -80 °C.
  Determinations of:
  - Serum bilirubin (mg/dL),
  will be carry out by dry chemistry using a Vitros 350 Analyzer.
Analysis of biochemicals variables (Aspartate amino transaminase) | 8 weeks
  Biochemical measurements at baseline and after 8 weeks supplementation Blood samples will be taken after 8 to 10 h of fasting and then centrifuged to obtain the serum, which will be frozen at -80 °C.
  Determinations of:
  - Aspartate amino transaminase (U/L),
  will be carry out by dry chemistry using a Vitros 350 Analyzer.
Analysis of biochemicals variables (Alanine amino transaminase) | 8 weeks
  Biochemical measurements at baseline and after 8 weeks supplementation Blood samples will be taken after 8 to 10 h of fasting and then centrifuged to obtain the serum, which will be frozen at -80 °C.
  Determinations of:
  - Alanine amino transaminase (U/L)
  will be carry out by dry chemistry using a Vitros 350 Analyzer.
Analysis of biochemicals variables (Gamma glutamyl transpeptidase) | 8 weeks
  Biochemical measurements at baseline and after 8 weeks supplementation Blood samples will be taken after 8 to 10 h of fasting and then centrifuged to obtain the serum, which will be frozen at -80 °C.
  Determinations of:
  - Gamma glutamyl transpeptidase (U/L),
  will be carry out by dry chemistry using a Vitros 350 Analyzer.
Analysis of biochemicals variables (Alkaline phosphatase) | 8 weeks
  Biochemical measurements at baseline and after 8 weeks supplementation Blood samples will be taken after 8 to 10 h of fasting and then centrifuged to obtain the serum, which will be frozen at -80 °C.
  Determinations of:
  - Alkaline phosphatase (U/L)
  will be carry out by dry chemistry using a Vitros 350 Analyzer.
Analysis of biochemicals variables (Urea) | 8 weeks
  Biochemical measurements at baseline and after 8 weeks supplementation Blood samples will be taken after 8 to 10 h of fasting and then centrifuged to obtain the serum, which will be frozen at -80 °C.
  Determinations of:
  - Urea (mg/dL)
  will be carry out by dry chemistry using a Vitros 350 Analyzer.

CONTACTS AND LOCATIONS:
Locations (2):
- Mexico (2):
  - University of Guadalajara, Guadalajara, Jaliscco
  - Universidad de Guadalajara, Guadalajara, Jalisco

REFERENCES:
- [Background] Basith S, Cui M, Hong S, Choi S. Harnessing the Therapeutic Potential of Capsaicin and Its Analogues in Pain and Other Diseases. Molecules. 2016 Jul 23;21(8):966. doi: 10.3390/molecules21080966. PMID 27455231
- [Background] Zheng J, Zheng S, Feng Q, Zhang Q, Xiao X. Dietary capsaicin and its anti-obesity potency: from mechanism to clinical implications. Biosci Rep. 2017 May 11;37(3):BSR20170286. doi: 10.1042/BSR20170286. Print 2017 Jun 30. PMID 28424369
- [Background] Joseph MSc A, John PhD F, Thomas MSc JV, Sivadasan SDP, Maliakel PhD B, Mohan PhD R, I M K. Influence of a Novel Food-Grade Formulation of Red Chili Extract (Capsicum annum) on Overweight Subjects: Randomized, Double-Blinded, Placebo-Controlled Study. J Diet Suppl. 2021;18(4):387-405. doi: 10.1080/19390211.2020.1780363. Epub 2020 Jun 24. PMID 32578488